CLINICAL TRIAL: NCT06780618
Title: The Effects of Brown Rice Consumption Compared to White Rice on Postprandial Changes in Interleukin-6 and Malondialdehyde Levels in Sedentary Workers
Brief Title: The Effects of Brown Rice Compared to White Rice on Postprandial Changes in IL-6 and MDA Levels in Sedentary Workers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Wulandari Taradita, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24-10-1628
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Sedentary Employees; Postprandial Oxidation and inﬂammation
Keywords: brown rice; white rice; interleukin-6; malondialdehyde; sedentary; inflammation; oxidative stress; postprandial
MeSH Terms: conditions — Sedentary Behavior; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- brown rice (Active Comparator)
  Interventions: Other: RICE
- white rice (Placebo Comparator)
  Interventions: Other: rice wheat (placebo)

INTERVENTIONS:
Other: RICE — 150 g of brown rice from Aek Sibundong variant at once
  Arms: brown rice
Other: rice wheat (placebo) — 150 g of white rice from Setra Ramos variant at once
  Arms: white rice

SUMMARY:
The goal of this clinical trial is to learn if brown rice and white rice affect oxidative stress and inflammation in office workers who don't exercise much. The main question it aims to answer is:

Does eating brown rice change MDA and IL-6 levels differently than eating white rice in people who don't exercise much?

Participants will:

Be interviewed to collect personal data, medical history, lifestyle habits, and dietary patterns.

Be measured to calculate Body Mass Index (BMI). Be interviewed to complete a questionnaire to assess their physical activity level in the past week.

Be interviewed to record all food and beverages consumed in the past 24 hours. Blood samples will be drawn twice, before and after consuming the research meal.

Be provided with a research meal consisting of rice (either brown or white), scrambled eggs, and tofu stew that must be finished within 15 to 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* healthy administrative employees,
* age 21-59 years,
* normal body mass index (18.5-22.9 kg/m2),
* low physical activity (≤600 METs minutes/week),
* assign for informed consent

Exclusion Criteria:

* being pregnant/breastfed/menopause,
* consumption of herbal medicines and/or supplements within 24 hours before data collection,
* having history of DM, CVD, cancer, and autoimmune disease,
* being vegan,
* smoking/alcohol drinking,
* allergic to research food's ingredients

Ages: 21 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
The Effects of Brown Rice Consumption Compared to White Rice on Postprandial Changes in Interleukin-6 and Malondialdehyde Levels in Sedentary Workers | Enrollment process to fullfil sample size at 2 weeks. The intervention will be completed in 1 day.

CONTACTS AND LOCATIONS:
Overall Officials: Wulandari Taradita, MD, Principal Investigator — Department of Nutrition Faculty of Medicine University of Indonesia
Locations (1):
- Faculty of Medicine University of Indonesia, Jakarta, Jakarta Special Capital Region, Indonesia